CLINICAL TRIAL: NCT06302114
Title: Upper Extremity Asymmetries in Overhead Athletes: Relationship With Injury and Performance
Brief Title: Upper Extremity Asymmetries in Overhead Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Research assistant, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Tubitak
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Extremity Asymmetries; Injury;Sports; Performance
Keywords: Asymmetry; Injury; Performance; Overhead
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes in overhead sports (Experimental): 15 years and older elite overhead athletes (swim, tennis, basketball,volleyball) were included in the study.
  Interventions: Other: Assessment of overhead athletes

INTERVENTIONS:
Other: Assessment of overhead athletes — Assessment of medicine ball forward throw, Y balance test, Range of motion of the shoulder (internal and external rotation), strength of internal and external rotator muscles.

SUMMARY:
Although overhead sports have different characteristics, the movements in the shoulder and upper extremity are similar. These sports may involve a combination of symmetrical, asymmetrical, bilateral and unilateral movements. In sports involving asymmetric movements, biomechanical changes are observed in that area due to the use of the dominant extremity. One of the reliable methods to reveal the stress effects caused by biomechanical stresses is to determine limb asymmetries. Considering the literature, limb asymmetries may be related to injury and performance.

ELIGIBILITY:
Inclusion Criteria:

* 15 years and older
* Attending regular sports training and competitions

Exclusion Criteria:

* Acute injury during tests

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Medicine ball forward throw | From enrollment to the end of assessment for 1 day
  The medicine ball forward throwing test is used to determine anaerobic power in athletes. The farthest distance the medicine ball is thrown from the starting position is recorded
Y balanced test | From enrollment to the end of assessment for 1 day
  Y balance test for the upper extremity is a test that evaluates the performance of the extremities and core balance. While one hand is fixed on the platform, the other hand tries to reach in the anterior, posterolateral and posteromedial directions. The furthest distance reached is recorded. The test is repeated for both extremities.
Range of motion of internal and external rotation | From enrollment to the end of assessment for 1 day
  While the athletes lie on their back, the shoulder is abducted at 90 degrees and the elbow is flexed at 90 degrees, internal and external rotation degrees are measured using a universal goniometer.
Strength of Internal and External Rotator Muscles | From enrollment to the end of assessment for 1 day
  While the athletes are lying on their back, with the shoulder in 90 degrees of abduction and the elbow in 90 degrees of flexion, internal and external rotation degrees are measured using the Commander Powertrack II dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Kızmaz, Principal Investigator — Munzur University; Fatma Ünver, Professor, Study Director — Pamukkale University; Pınar Toksöz, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Pamukkale, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No